CLINICAL TRIAL: NCT00343590
Title: Whole Body Vibration Therapy in a Participant With Multiple Sclerosis Related Balance Deficits - A Case Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCC-06-03
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

INTERVENTIONS:
Device: Whole Body Vibration machine

SUMMARY:
The purpose of this investigation is to determine the effect of Whole Body Vibration Therapy (WBV) on balance in a participant with multiple sclerosis (MS) related balance deficits as measured by the NeuroCom Balance Master, the Sapphire IIME EMG Device and the Kurtzke Expanded Disability Status Scale (EDSS) and the Berg Balance Score.

ELIGIBILITY:
Inclusion Criteria:

Logan student, staff, or faculty or general public with a minimal of 2 year history of diagnosed Multiple Sclerosis (MS)

Exclusion Criteria:

1)visual or vestibular condition that would affect balance; 2) Non-Ms related systemic illness that would have an adverse effect on balance; 3) Local infection, acute inflammation, injury, tumors or other malignancy, recent wounds, diabetes; 4) Any unstable joints of the lower extremity, recent hip and knee joints or fitted hip or knee pins, bolts and/or plates; 5) Acute thrombosis; 6) Severe migraine, epilepsy; 7) Serious cardiovascular disease, wearing a pacemaker; Any Spinal manipulation within 48 hours; 8) Acute disc herniation, discopathy or spondylolysis; 9) Prescription or herbal muscle stimulants, relaxants, etc. that could affect balance; 10) Any implanted device or prosthesis or intrauterine IUD type of device; 11) Pregnancy

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
NeuroCom Balance Master
SF-EMG Nerve conduction velocity test
Berg balance score

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Enix, DC, Principal Investigator — Logan College of Chiropractic
Locations (2):
- United States (2):
  - Logan College of Chiropractic, Chesterfield, Missouri
  - Logan College of Chirpractic, Chesterfield, Missouri

REFERENCES:
- [Background] Romberg A, Virtanen A, Ruutiainen J, Aunola S, Karppi SL, Vaara M, Surakka J, Pohjolainen T, Seppanen A. Effects of a 6-month exercise program on patients with multiple sclerosis: a randomized study. Neurology. 2004 Dec 14;63(11):2034-8. doi: 10.1212/01.wnl.0000145761.38400.65. PMID 15596746
- [Background] Griffin JW. Use of proprioceptive stimuli in therapeutic exercise. Phys Ther. 1974 Oct;54(10):1072-9. doi: 10.1093/ptj/54.10.1072. No abstract available. PMID 4422763